CLINICAL TRIAL: NCT06816576
Title: Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University
Brief Title: The Effect of Emotional Freedom Techniques Application on Patients With Cancer Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: okutan1
Record Dates: First submitted 2025-02-02; First posted 2025-02-10 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Complications; Emotion Regulation; Death Anxiety
Keywords: Death Anxiety; postoperative; Emotional Freedom Technique; cancer phobia
MeSH Terms: conditions — Postoperative Complications; Emotional Regulation; Necrophobia; Pathophobia

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pre-testpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After coming to the clinic after surgery and after their condition was stable, the patients were given the patient introduction form, subjective discomfort unit, cancer anxiety scale and death anxiety scale as a pre-test. The researchers provided EFT training to the patients and asked them to apply EFT. After an average of 3 days, the subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a post-test.
  Interventions: Other: Emotional Freedom Technique
- Control Group (No Intervention): After coming to the clinic after surgery and after their condition was stable, the patient introduction form, subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a pre-test. No intervention was made to the control group patients outside the clinical protocol. After an average of 3 days, the subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a post-test.

INTERVENTIONS:
Other: Emotional Freedom Technique — Emotional Freedom Technique application; It is an application that works on cognitive and energetic levels. Emotional Freedom Technique Application Instructions
  1. Determination of Subjective Units of Disturbance (SUD)
  2. Preparation or setup
  3. Application of appropriate acupuncture points in order
  4. 9-Gamut: An application that allows the two hemispheres of the brain to be stimulated simultaneously
  5. Application of appropriate acupuncture points in order again
  6. Control of the differentiation in the level of discomfort with Subjective Units of Disturbance again
  Arms: Intervention Group

SUMMARY:
The aim is to examine the effect of Emotional Freedom Technique on death anxiety in patients with postoperative cancer phobia.

The hypotheses of the study are as follows:

H0: Emotional Freedom Technique has no effect on postoperative death anxiety in patients with cancer phobia.

H1: Emotional Freedom Technique has a positive effect on postoperative death anxiety in patients with cancer phobia.

DETAILED DESCRIPTION:
Intervention Group

After coming to the clinic after surgery and after their condition was stable, the patients were given the patient introduction form, subjective discomfort unit, cancer anxiety scale and death anxiety scale as a pre-test. The researchers provided Emotional Freedom Technique (EFT) training to the patients and asked them to apply Emotional Freedom Technique. After an average of 3 days, the subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a post-test.

Control Group

After coming to the clinic after surgery and after their condition was stable, the patient introduction form, subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a pre-test. No intervention was made to the control group patients outside the clinical protocol. After an average of 3 days, the subjective discomfort unit, cancer anxiety scale and death anxiety scale were applied as a post-test.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Having had oncological surgery,
* Having no visual or auditory problems,
* Having no psychiatric problems.

Exclusion Criteria:

* Not accepting to participate in the study or wanting to leave,
* Being under 18 years of age,
* Having been previously diagnosed with cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
death anxiety | After coming to the clinic after surgery and their condition becoming stable, the death anxiety scale was applied to the patients as a pre-test. Three days later, the death anxiety scale was applied as a post-test.
  Death Anxiety Scale:
  The scale developed by Templer was translated into Turkish by Sarıkaya and Baloğlu. The scale consists of 20 items. High scores indicate high death anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, Dr., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)